CLINICAL TRIAL: NCT02019875
Title: Effect of Modulating CYP3A4 Activity on Mineral Homeostasis
Brief Title: CYP3A4 Activity and Mineral Homeostasis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Thummel, Professor, Department of Pharmaceutics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001894; R01GM063666 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D and Calcium Homeostasis
Keywords: Vitamin D; CYP3A4; Calcium
MeSH Terms: interventions — Rifampin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Water (Placebo Comparator): 200 mL of water once a day for 14 days
  Interventions: Other: Placebo
- Rifampin (Active Comparator): Rifampin 600 mg once a day for 14 days
  Interventions: Drug: Rifampin
- Grapefruit Juice (Active Comparator): 200 mL of grapefruit juice once a day for 14 days
  Interventions: Other: Grapefruit Juice
- Grapefruit Juice Plus Rifampin (Active Comparator): 200 mL of grapefruit juice once a day for 8 days plus rifampin 600 mg once a day for 14 days
  Interventions: Drug: Rifampin; Other: Grapefruit Juice
- Clarithromycin (Active Comparator): Clarithromycin 250 mg twice a day for 14 days
  Interventions: Drug: Clarithromycin
- Clarithromycin Plus Rifampin (Active Comparator): Clarithromycin 250 mg twice a day for 14 days plus rifampin 600 mg once a day for 14 days
  Interventions: Drug: Rifampin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Rifampin — P450 inducer
  Other Names: Rifadin
  Arms: Clarithromycin Plus Rifampin; Grapefruit Juice Plus Rifampin; Rifampin
Drug: Clarithromycin — CYP3A4 and Pgp inhibitor in both intestine and liiver
  Other Names: Biaxin
  Arms: Clarithromycin; Clarithromycin Plus Rifampin
Other: Grapefruit Juice — CYP3A4 inhibitor in intestine
  Arms: Grapefruit Juice; Grapefruit Juice Plus Rifampin
Other: Placebo
  Arms: Water

SUMMARY:
The purpose of this study is to determine whether changes in the activity of the enzyme CYP3A4 can change the Vitamin D and bone mineral homeostasis.

DETAILED DESCRIPTION:
Healthy volunteers will receive one of six interventions for 14 days (determined by randomization):a). 200 mL of water once a day; b) rifampin 600 mg once a day; c) 200 mL of grapefruit juice once a day for 8 days plus rifampin 600 mg once a day for 14 days; d) clarithromycin 250 mg twice a day; f) clarithromycin 250 mg twice a day plus rifampin 600 mg once a day.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no history of significant medical conditions including cardiac, pulmonary, gastrointestinal, or renal disease, HIV, diabetes mellitus or Hepatitis B or C
* Subjects will be males or females 18-60 years of age
* Subjects must read and understand English
* Subjects must be able to provide informed consent
* Subjects must be willing to avoid prescription medications, OTC drugs, dietary supplements and foods that are known to modulate CYP3A4 expression or activity
* Subjects must be willing to maintain a consistent consumption of calcium and Vitamin D during the study and maintain a daily logbook of their dietary consumption
* Women not currently pregnant or lactating. In addition, women participants of childbearing age must be willing to utilize a barrier method of birth control (sterilization will be acceptable)
* Subjects will have no known allergies to the study drugs to be used
* Subject's corrected QTc interval obtained by electrocardiogram will be ≤ 430 ms in men or ≤ 450 ms in women

Exclusion Criteria:

* Subjects with any significant chronic medical condition, including cardiac, pulmonary, gastrointestinal, or renal disease, HIV, diabetes mellitus or Hepatitis B or C
* Subjects less than 18 or greater than 60 years of age
* Subjects unable to read and understand English
* Subjects unable to provide informed consent
* Subjects unable to avoid prescription medications, OTC drugs, dietary supplements and foods that are known to modulate CYP3A4 expression or activity
* Subjects not willing to maintain a consistent consumption of calcium and Vitamin D during the study and maintain a daily logbook of their dietary consumption
* Women who are pregnant or lactating and women participants of childbearing age not willing to utilize a barrier method of birth control (sterilization will be acceptable)
* Subjects with allergies to rifampin, clarithromycin or grapefruit juice
* Potential participants will be excluded if they are concurrently participating in another research study
* Subjects with corrected QTc interval > 430 ms in men or > 450 ms in women on electrocardiogram

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Thummel, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Water: 200 mL of water once a day for 14 days
  Placebo
Period: Overall Study
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Started | 16 | 18 | 15 | 15 | 16 | 12
Completed | 14 | 16 | 15 | 14 | 15 | 11
Not Completed | 2 | 2 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin | Total
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.6) | 29.5 (8.3) | 32.1 (11.1) | 29.9 (9.1) | 28.1 (9.3) | 27.3 (8.0) | 29.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 13 | 10 | 9 | 5 | 51
  Male | 6 | 10 | 2 | 4 | 6 | 6 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Not Hispanic or Latino | 14 | 15 | 14 | 14 | 15 | 9 | 81
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 3 | 4 | 4 | 4 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 2 | 0 | 0 | 1 | 0 | 4
  White | 10 | 11 | 11 | 9 | 10 | 11 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 1, 25(OH) D3 Vitamin D
Description: Serum 1, 25(OH) D3 Vitamin D
Time Frame: Samples will be collected on days 1, 4 and 7, and day 22 (last day of intervention). Treatment began on day 8. Data presented is day 22 concentration - Baseline (the average of day 1, day 4 and day 7 concentrations).
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: pM
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
pM | 3.2 [-11 to 17.4] | 1.7 [-12 to 15.4] | 3.7 [-10.5 to 17.9] | -3.3 [-17.5 to 10.9] | -4.7 [-18.4 to 9.0] | 0.4 [-15.7 to 16.4]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.884, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-21.2 to 18.3]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.955, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-19.5 to 20.7]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-26.5 to 13.6]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.434, Mixed Models Analysis; Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-27.6 to 11.9]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.796, Mixed Models Analysis; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-24.2 to 18.6]

2. Primary Outcome: 25(OH) D3 Vitamin D
Description: Serum 25(OH) D3 Vitamin D
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: nM
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
nM | -3.1 [-6.6 to 0.4] | -4.3 [-7.7 to -1.0] | -1.3 [-4.8 to 2.1] | -1.6 [-5.1 to 1.8] | 0.6 [-2.8 to 3.9] | -5.0 [-8.9 to -1.1]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-6.0 to 3.6]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.482, Mixed Models Analysis; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-3.1 to 6.7]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.559, Mixed Models Analysis; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-3.4 to 6.4]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.138, Mixed Models Analysis; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-1.2 to 8.5]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.477, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-7.1 to 3.3]

3. Primary Outcome: Parathyroid Hormone
Description: Blood Parathyroid Hormone
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
pg/mL | 0.3 [-7.9 to 8.4] | 0.4 [-7.2 to 8.1] | 1.6 [-6.3 to 9.5] | 1.0 [-7.2 to 9.1] | 2.7 [-5.2 to 10.6] | 0.6 [-8.6 to 9.8]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.98, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-11.0 to 11.3]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-10.0 to 12.7]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-10.8 to 12.2]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-8.9 to 13.8]
Statistical Analysis 5: Comparison: Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-11.9 to 12.6]

4. Primary Outcome: Osteocalcin
Description: Serum Osteocalcin
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
ng/mL | 0.0 [-1.1 to 1.2] | -1.1 [-2.2 to 0.0] | 0.7 [-0.5 to 1.8] | 0.0 [-1.2 to 1.1] | 3.7 [2.6 to 4.8] | 4.0 [2.7 to 5.2]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.7 to 0.5]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.44, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.0 to 2.2]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.7 to 1.6]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [2.1 to 5.2]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [2.2 to 5.6]

5. Primary Outcome: Calcium, Ionized
Description: Serum
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
mM | 0.0 [-0.014 to 0.014] | -0.008 [-0.021 to 0.005] | -0.017 [-0.031 to -0.003] | -0.011 [-0.025 to 0.003] | -0.005 [-0.019 to 0.008] | -0.009 [-0.025 to 0.008]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.027 to 0.012]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = -0.017, 95% CI 2-sided [-0.037 to 0.003]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Final Values) = -0.011, 95% CI 2-sided [-0.031 to 0.009]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.025 to 0.015]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.03 to 0.014]

6. Primary Outcome: Calcium/Creatinine (mg/g)
Description: Urine Calcium/Creatinine (mg/g)
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: ratio (mg/g)
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
ratio (mg/g) | 3.4 [-24.9 to 31.8] | -9.2 [-36.5 to 18.2] | -41.1 [-69.4 to -12.7] | -3.8 [-32.1 to 24.5] | 6.3 [-21.1 to 33.6] | 41.4 [9.5 to 73.3]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-52.0 to 26.7]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.03, Mixed Models Analysis; Mean Difference (Final Values) = -44.5, 95% CI 2-sided [-84.5 to -4.5]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-47.3 to 32.8]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-36.6 to 42.2]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.08, Mixed Models Analysis; Mean Difference (Final Values) = 38.0, 95% CI 2-sided [-4.7 to 80.6]

7. Primary Outcome: Phosphate/Creatinine (mg/g)
Description: Urine Phosphate/Creatinine(mg/g)
Time Frame: as for outcome 1
Population: Comparison of treatment effect (end of treatment - baseline) between treatment groups.
Measure: Mean (95% Confidence Interval); unit: ratio (mg/g)
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
Number analyzed (Participants) | 14 | 16 | 15 | 14 | 15 | 11
ratio (mg/g) | 8.3 [-69.0 to 85.5] | 11.1 [-63.5 to 85.7] | 23.3 [-54.0 to 100.5] | 79.6 [2.3 to 156.8] | 5.5 [-69.1 to 80.1] | 60.0 [-27.1 to 147.1]
Statistical Analysis 1: Comparison: Water vs Rifampin; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-104.5 to 110.2]
Statistical Analysis 2: Comparison: Water vs Grapefruit Juice; Test type: Superiority; p = 0.79, Mixed Models Analysis; Mean Difference (Final Values) = 15.0, 95% CI 2-sided [-94.2 to 124.2]
Statistical Analysis 3: Comparison: Water vs Grapefruit Juice Plus Rifampin; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = 71.3, 95% CI 2-sided [-37.9 to 180.5]
Statistical Analysis 4: Comparison: Water vs Clarithromycin; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-110.1 to 104.7]
Statistical Analysis 5: Comparison: Water vs Clarithromycin Plus Rifampin; Test type: Superiority; p = 0.38, Mixed Models Analysis; Mean Difference (Final Values) = 51.8, 95% CI 2-sided [-64.7 to 168.2]

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Water | Rifampin | Grapefruit Juice | Grapefruit Juice Plus Rifampin | Clarithromycin | Clarithromycin Plus Rifampin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/15 | 0/15 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18 | 0/15 | 0/15 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 1/16 | 1/18 | 0/15 | 1/15 | 0/16 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water (N=16) | Rifampin (N=18) | Grapefruit Juice (N=15) | Grapefruit Juice Plus Rifampin (N=15) | Clarithromycin (N=16) | Clarithromycin Plus Rifampin (N=12)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | NA | 1 (1)
elevated transaminase (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
None noted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT02019875/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT02019875/SAP_001.pdf